CLINICAL TRIAL: NCT04793035
Title: An Observational Clinical Feasibility Study of the Omega Cuff Device for GERD
Brief Title: Omega Cuff for GERD Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aplos Medical (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-0001-000
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: GERD, Acid Reflux, Treatment
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: The study is an observational, prospective, non-randomized, open-label, feasibility study of patients receiving the Ω-Cuff device. The study is intended to evaluate the safety of the Ω-Cuff device and its ability to reduce the symptoms of GERD by augmenting the function of the LES. The study will be performed at up to three (3) investigational centers in the US with a maximum of 15 subjects who will be implanted with the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Enrolled patients (Experimental): Single-arm study for enrolled GERD patients to be treated with an Omega-Cuff device
  Interventions: Device: Omega-Cuff

INTERVENTIONS:
Device: Omega-Cuff — An omega-shaped nitinol device to be placed and secured on the Lower Esophageal Sphincter area

SUMMARY:
This clinical feasibility study is to evaluate the performance of the Omega-Cuff in the treatment of acid reflux for up to 15 patients with a 1-year follow-up period. The Omega-shaped nitinol device is placed on top of the esophageal sphincter muscle just above the stomach in a laparoscopic surgical procedure without altering anatomy. In animal studies, the device safely increased the pressure on the sphincter, meaning it increased resistance to acid reflux, but did not interfere with normal food swallowing, meaning food went down to the stomach normally and smoothly. The device is intended to augment the function of the weak sphincter in minimizing acid reflux but allows easy swallowing of food in GERD patients. The clinical feasibility study is to see how well this device functions in patients and to assess its safety profile. This is a permanent implant that will last the lifetime of the patient. The device will not interfere with patients who may need diagnostic MRI scans. The device can be safely removed if needed.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease (GERD) is a chronic excessive stomach content reflux that results in heartburn with major adverse impacts on patient quality of life. It is increasingly common in industrialized societies with a prevalence of ~7% of the population experiencing symptoms daily.

A weak Lower Esophageal Sphincter allows excessive acidic stomach content to enter the esophagus. Drug is the most common GERD symptoms relief. Proton pump inhibitors (PPI's) drugs, such as Prevacid® reduce stomach acid production but not reflux. PPIs fail to treat 10% to 20% of the patients. Up to 40% of patients become refractive in long-term use and develop serious side effects.

The next level treatments are surgeries, i.e., Nissen Fundoplication, the LINX® Magnetic Esophageal Sphincter. Both Nissen and LINX are effective but have many aggravating side effects including dysphagia, gas, bloating, increased flatus, difficulty with belching, or vomiting, device erosion and removal, MRI incompatibility, and reoperations.

Omega-Cuff The Omega-Cuff device augments the LES as a partial fundoplication but without stomach involvement. The Ω-shaped scaffold structure is placed around the outside of the esophagus to help the weak LES restoring its barrier function. When swallowing, the Ω-Cuff, along with the uncovered esophageal tissue, smoothly expands to allow food passage. It provides resistance to gastric reflux yet allows easy swallowing.

The rationale for this early feasibility trial is to establish a basic safety profile and refine the implant technique to support a pivotal clinical trial (via an IDE supplement). Evaluating its performance characteristics will better define the efficacy requirements for the pivotal trial.

The single-use Omega-Cuff device is a one-piece, Ω-shaped scaffold structure. It is placed at the LES region through an open incision or through a laparoscopic port with a minimum internal diameter of 15mm. Five device sizes, 14-20 mm (nominal) in diameter, are available to accommodate varying patient anatomy. It has attachment sites for sutures attachment at the top and bottom end of the device to the esophagus.

The esophagus circumference is measured with a suture or tape and converts into the esophagus diameter. A table shows the size of the device to use based on the esophagus diameter. When the measured length is between sizes, use the next smaller device size.

If the Omega Cuff is unable to be placed for any reason, a standard of care surgical treatment can be offered to the patient or the patient may elect to have the surgery aborted.

The Omega-Cuff device is indicated for patients diagnosed with GERD, as defined by abnormal pH testing, and who continue to have chronic GERD symptoms despite maximum medical therapy for the treatment of reflux.

The study is a prospective, non-randomized, open-label feasibility study of patients receiving the Ω-Cuff device. The study intends to evaluate the safety of the Ω-Cuff and its ability to reduce the symptoms of GERD by augmenting the function of the LES. The study will be performed at up to 3 investigational sites in the US and a maximum of 15 subjects ages 22-74 to be implanted with the device. The information from this study will be used to support the design and conduct of a pivotal clinical trial.

The study will follow the standard clinical trial practices of Informed Consent (including HIPAA authorization), screening, Safety Measurements, Adverse Events and reporting, follow-up assessments at discharge, 2-4 weeks, 2, 3, 6, 9, and 12 months minimum post-procedure visits. Depending on the follow-up period, predetermined items will be performed and recorded. These include a chest/abdominal X-ray to ensure the device remains correctly placed, any adverse events, completing the GERD-HRQL form and 24-hr pH profile with the subject discontinued any PPI therapy or anti-reflux medication for at least 10 days, manometry, endoscopy, barium esophagram, and health history.

Because of the small sample size, there are no statistically derived endpoints for this feasibility study. The primary safety parameter will be the rate of all adverse events at various time points. The effectiveness endpoint of this study will be based on normalization of pH (with normalization defined as pH <4 for no more than 4.5% of monitoring time) or reduction of at least 50% in total time that pH <4, relative to baseline. Another endpoint will be at least a 50% improvement in the GERD-HRQL scores at 12 months, and the reduction of daily PPI use by subjective measurements using the GERD-HRQL, and LES function will be characterized by objective measurements using 24hr pH profile, manometry/motility, endoscopy, and barium esophagram. The Ω-Cuff can be surgically removed if there are serious issues with the device. Depending on the circumstances, the procedure could be laparoscopic, endoscopic, or laparotomic.

Data Analysis. This study is to develop an information set that will help the development of a pivotal clinical study plan. Experience implanting the study device in 15 subjects should be adequate for the investigator(s) to feel comfortable enough with the implant procedure to be able to teach it to other investigators in a pivotal clinical trial and to provide clear written direction in the Instructions for Use. Their experience and observations should also help elucidate any safety concerns that must be addressed before implementing a pivotal clinical trial. The demographic and baseline variables of interest will be summarized via standard descriptive statistics. As this is a single-arm trial, hypothesis testing is not possible on these variables. Results from summary statistics will be used in conjunction with available literature to provide sample size estimates for efficacy endpoints for a pivotal clinical trial.

Risk Analysis Conclusion. Ω-Cuff meets applicable principles of risk management, design control provisions of 21 CFR 820.3, and current standards. This study is not anticipated to pose new types of risks from those identified for similar products/procedures. To date, there is no evidence to suggest that the incidence of complications associated with the use of Ω-Cuff will be greater than the risks posed by other existing marketed products. Therefore, the likely benefit of the Ω-Cuff treatment in this controlled setting outweighs the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* • Subject must be at least 22 years of age and must be less than 75 years of age with a life expectancy > 3 years.

  * Subject is a suitable surgical candidate, i.e., is able to undergo general anesthesia and laparoscopic surgery.
  * Subject has documented typical symptoms of gastroesophageal reflux disease (GERD) for longer than 6 months (regurgitation or heartburn that is defined as a burning epigastric or substernal pain that responds to acid neutralization or suppression).
  * Subject requires daily proton pump inhibitor or other anti-reflux drug therapy.
  * Total Distal Ambulatory Esophageal pH must meet the following criteria: pH< 4 for ≥ 4.5% of the time Note: Subjects will have discontinued any GERD medications for at least 10 days prior to testing.
  * Subject has a symptomatic improvement on proton-pump inhibitor (PPI) therapy demonstrated by a GERD-Health-Related Quality of Life (GERD-HRQL) score of ≤ 10 on proton-pump inhibitors and ≥ 15 off PPIs, or subjects with a ≥ 6-point improvement when comparing his/her on-PPI and off-PPI GERD-HRQL score.
  * Subject has GERD symptoms in absence of PPI therapy (minimum 10 days).
  * If the subject is of child-bearing potential, she must have a negative pregnancy test within one week prior to implant and must agree to use effective means of birth control during the course of the study.
  * Subject is willing and able to cooperate with follow-up examinations.
  * Subject has been informed of the study procedures and the treatment and has signed an informed consent form.

Exclusion Criteria:

* • The procedure is an emergency procedure.

  * Subject is currently being treated with another investigational drug or investigational device.
  * Subject has a history of gastroesophageal surgery, anti-reflux procedures, or gastroesophageal/gastric cancer.
  * Subject has undergone any previous endoscopic anti-reflux intervention for GERD.
  * Subject has suspected or confirmed esophageal or gastric cancer.
  * Subject has any size hiatal hernia >3cm as determined by endoscopy.
  * Distal esophageal motility (average of sensors 3 and 4) is less than 35 mmHg peristaltic amplitude on wet swallows or <70% (propulsive) peristaltic sequences.
  * Subject has esophagitis Grade C or D (LA Classification).
  * Subject has a Body Mass Index (BMI)>35.
  * Subject has symptoms of dysphagia more than once per week within the last 3 months.
  * Subject is diagnosed with Scleroderma or an esophageal motility disorder such as but not limited to Achalasia, Nutcracker Esophagus, or Diffuse Esophageal Spasm or Hypertensive LES.
  * Subject has a history of or known esophageal stricture or gross esophageal anatomic abnormalities (Schatzki's ring, obstructive lesions, etc.).
  * Subject has esophageal or gastric varices.
  * Subject has a history of or known Barrett's esophagus.
  * Subject cannot understand trial requirements or is unable to comply with the follow-up schedule.
  * Subject is pregnant or nursing or plans to become pregnant during the course of the study.
  * Subject has a medical illness (e.g., congestive heart failure) that may cause the subject to be non-compliant with or unable to meet the protocol requirements or is associated with limited life expectancy (i.e., less than 3 years).
  * Subject is diagnosed with a psychiatric disorder (e.g., bipolar, schizophrenia, etc.); however, subjects who exhibit depression but are on appropriate medication(s) may be included.
  * Subject has suspected or known allergies to titanium, stainless steel, nickel, or ferrous materials.
  * Subject has an electrical implant or metallic abdominal implants.
  * Subject is not a surgical candidate for open laparotomy.

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | 12 months
  The primary safety parameter will be a summary at 12 months of the rate of all adverse events at various time points post-implant procedure. This will be compared to other GERD treatment results.
Outcome 2 | 12 months
  The primary effectiveness endpoint of this study is the pH measurements result. Efficacy here is defined as the amount of time the pH<4 is 4.5% of the time or less, or the amount of time with pH<4 is at least 50% less than the baseline measurement.
Outcome 3 | 12 months
  The primary quality of life endpoint will be at least a 50% improvement in the GERD-HRQL scores at 12 months.
Outcome 4 | 12 mohths
  Reduction of PPI usage. The reduction of daily PPI use by subjective assessment using the GERD-HRQL.
Outcome 5 | 12 months
  LES function. The LES function will be characterized by objective measurements using a 24hr pH profile, manometry/motility, endoscopy, and barium esophagram.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - HonorHealth, Scottsdale, Arizona
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No